CLINICAL TRIAL: NCT00540774
Title: Optical Sensor for Photodynamic Detection of Oral Pathology
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The PRMC committee has made the decision there is sufficient data to complete an analysis and publish findings.
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Livionex Inc. (Industry); Orahealth (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Petra E. Wilder-Smith, Professor of Surgery and Director of Dentistry, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20022805; R44CA265514 (NIH); T31IR1825 (Other Grant/Funding Number: California Tobacco-Related Diseases Research Program); R03EB014852 (NIH); R01DE022831 (NIH); LDG (Other: Livionex); OE (Other: Oral Essentials); UCI-08-52 (Other: UCI Chao Family Comprehensive Cancer Center)
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Mouth Diseases
Keywords: Oral cancer; Oral mucositis; Periodontitis; Dry mouth; Gingivitis; Oral lesions; Dental Hard Tissues; Oral Biofilm
MeSH Terms: conditions — Mouth Diseases; Mouth Neoplasms; Stomatitis; Periodontitis; Xerostomia; Gingivitis

STUDY DESIGN:
Masking Description: No masking other than an anonymization of data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral tissue (Other): Imaging of oral structures and pathologies
  Interventions: Device: detection of oral pathology

INTERVENTIONS:
Device: detection of oral pathology — detection of oral pathology

SUMMARY:
Overall objective of this work is to develop better ways of detecting, diagnosing and measuring oral diseases and structures using light and optical approaches. All different areas of the mouth will be imaged, including healthy, diseased, dysplastic and malignant, as well as oral biofilm, and the imaging data compared against conventional diagnostic approaches such clinical and histopathological and molecular evaluations to (1) gain a better understanding of processes involved in oral pathology and (2) develop a combined patient specific, non-invasive method for the detection, diagnosis and screening of oral pathology and biofilm. Thus our goal is to identify and evaluate microstructural, metabolic, vascular, protein, genomic and metabolomics biomarkers of oral pathology can be used to detect, predict and map oral pathology, especially neoplasia.

We are recruiting patients with a wide range of oral conditions including plaque, dry mouth, toothache, root canal treatments, gum disease, oral sores, dysplasia and cancer, autoimmune conditions and others as well as healthy control subjects. We will use a range of non-invasive imaging modalities to obtain information on the ways in which the oral health status affects optical properties, and determine means of detecting and quantifying these factors.. Imaging modalities to be utilized include:

1. Coherence and Doppler Tomography
2. Laser Speckle Imaging
3. Various forms of Spectroscopy
4. Fluorescence

DETAILED DESCRIPTION:
Purpose of the research is to identify optical predictors and biomarkers of health and disease.

Hypothesis: microstructural, metabolic, vascular, protein, genomic and metabolomics biomarkers of oral pathology can be used to detect, predict and map oral pathology, especially neoplasia.

Researchers of the Beckman Laser Institute (BLI) have developed many non-invasive imaging modalities for assessment of oral tissue. This protocol will allow data acquisition with these multiple modalities to allow validation of data. Imaging modalities to be utilized include:

1. Coherence and Doppler Tomography (OCT)
2. Laser Speckle Imaging (LSI)
3. Photon Migration Spectroscopy (PMS)
4. Autofluorescence Imaging

In addition, saliva samples from the patients will be analyzed and the resulting data regarding the dysregulation in the activities of genes, proteins and other molecules will be correlated with findings from different imaging systems with respect to the stage of oral carcinogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18 years and older
* Have oral lesion or not have oral lesion
* Have condition of dry mouth
* Have condition of Gum disease
* Non-smoker

Exclusion Criteria:

* Age less than 18 years old
* Advanced gum disease, diseases of oral tissue
* Untreated cavities
* Pregnant or breastfeeding
* Immune compromised individuals

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2003-04; Primary Completion 2025-06-03 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Healthy oral tissue | up to 12 months
  Develop a non-invasive tool for the detection, diagnosis and screening of oral pathology and understanding of processes involved in oral pathology

CONTACTS AND LOCATIONS:
Overall Officials: Petra Wilder-Smith, DDS, PhD, Principal Investigator — University of Calfornia Irvine
Locations (1):
- Beckman Laser Institute and Medical Clinic, Irvine, California, United States